CLINICAL TRIAL: NCT05408897
Title: Prediction of Postoperative Treatment Efficacy and Recurrence Risk of High-risk GIST Based on Minimal Residual Disease Detected by Liquid Biopsy
Brief Title: Prediction of Postoperative Treatment Efficacy and Recurrence Risk of High-risk GIST Based on Liquid Biopsy MRD
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, YE Yingjiang, Director of the department of gastrointestinal surgery, Peking University People's Hospital
Other Study IDs: WCJZL202103
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Stromal Tumors; Minimal Residual Disease
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm, Residual | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissues: collected from preoperative needle biopsy or specimens of surgical resection
  blood tissues: venous blood collected at specific time point stipulated in the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liquid biopsy — A test that enables the diagnosis or analysis of tumors using only a blood or fluid sample rather than a solid tissue biopsy.

SUMMARY:
So far, MRD assessment by liquid biopsy (ctDNA) has not been used to predict postoperative treatment efficacy and recurrence risk of GIST patients because of special disease characteristics and technological limitations. Therefore, we conducted this prospective multi-center, single-arm observational study to collect 45 operable patients with locally advanced, suspected high-risk GIST. NGS genetic testing platform is used to detect tumour tissues and peripheral ctDNA will also be dectected. we try to explore the correlation between PFS/OS and MRD in high-risk GIST patients by analyzing the relationship between dynamic changes in ctDNA mutation spectrum and postoperative adjuvant therapy efficacy, and to evaluate MRD-based genomic characteristics to guide further treatment.

DETAILED DESCRIPTION:
Assessing MRD (Minimal Residual Disease) and predicting the postoperative adjuvant treatment efficacy and recurrence risk of tumor patients based on ctDNA (circulating tumor DNA) detected by liquid biopsy have been exploratorily studied and applied in many types of cancers. However, as for GISTs (gastrointestinal stromal tumors), the most common mesenchymal neoplasm of the gastrointestinal tract, they have less peripheral ctDNA fragments compared with those tumors of hematological or epithelial origins. Since there are also some limitations of previous detection technology and detection depth, prospective study for prediction of postoperative treatment efficacy and recurrence risk of high-risk GIST is lacking.

In this study, a prospective multi-center, single-arm observational study is conducted to collect operable patients with locally advanced GIST. According to results of preoperative imaging examinations or pathological biopsy, 45 high-risk GIST patients will be screened and enrolled. Next-Generation Sequencing (NGS) genetic testing platform (Burning Rock Oncoscreen Plus TM) is used to detect the baseline tumour tissues (detection depth 1000X) of these patients. And peripheral ctDNA (detection depth 30000X) of multiple pre/postoperative time points will be detected. The genetic profile and clinical information of each patient will be collected. Combining all the information, bioinformatics analysis will be carried out on the gene detection results of these patients at each time point, and the correlation between the postoperative recurrence time and the ctDNA positive rate/postoperative clearance rate of patients will be compared. The characteristics changes and dynamic changes of tumor release degree will also be analyzed. To explore the correlation between PFS/OS and MRD in high-risk GIST patients, we plan to analyze the relationship between dynamic changes in ctDNA mutation spectrum and postoperative adjuvant therapy efficacy, and to evaluate MRD-based genomic characteristics to guide further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80
* Patients suspected for high-risk GIST by preoperative imaging examinations or diagnosed with high-risk GIST by pathological biopsy, who have not received preoperative neoadjuvant treatment
* Patients must have not received any treatment including radiotherapy, chemotherapy or surgery
* The function of other organs including liver and kidneys is good enough so that the patients could tolerate targeted therapy and surgery
* Postoperative pathology conformed the diagnosis of high-risk GIST
* Patients and their families could understand the protocol of this study and voluntarily agree to participate in. Signed informed consents are required

Exclusion Criteria:

* Previous medical history of malignant tumors or synchronous other malignancies
* Emergent surgery because of bowel obstruction, perforation or bleeding
* Pregnant or lactant women
* Medical history of severe mental illness
* Patients with contraindication for targeted therapy and surgery
* Non-R0 resection
* Postoperative pathology conformed the diagnosis of non-high-risk GIST
* Patients with distant metastasis
* Other situations in which researchers consider that the patient is unsuitable for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study plans to invite patients with the following criteria: patients with resectable locally advanced GIST who received or did not receive neoadjuvant molecular targeted therapy, and patients with high recurrence risk grading by postoperative pathological assessment, including but not limited to the following clinical factors: Tumor Location, size, degree of mitoses, degree of tumor rupture, etc. Those who did not reach R0 resection or did not match the pathological staging, or who could not complete the test items required by the trial within the specified time due to the patient's non-cooperation, or who were deemed unsuitable by other investigators, would not be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
recurrence | 3 to 5 years
  Recurrence or metastasis of high-risk GIST after surgical resection followed by targeted drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Connolly EM, Gaffney E, Reynolds JV. Gastrointestinal stromal tumours. Br J Surg. 2003 Oct;90(10):1178-86. doi: 10.1002/bjs.4352. PMID 14515284
- [Result] Tran T, Davila JA, El-Serag HB. The epidemiology of malignant gastrointestinal stromal tumors: an analysis of 1,458 cases from 1992 to 2000. Am J Gastroenterol. 2005 Jan;100(1):162-8. doi: 10.1111/j.1572-0241.2005.40709.x. PMID 15654796
- [Result] Graadt van Roggen JF, van Velthuysen ML, Hogendoorn PC. The histopathological differential diagnosis of gastrointestinal stromal tumours. J Clin Pathol. 2001 Feb;54(2):96-102. doi: 10.1136/jcp.54.2.96. PMID 11215292
- [Result] Chan JK. Mesenchymal tumors of the gastrointestinal tract: a paradise for acronyms (STUMP, GIST, GANT, and now GIPACT), implication of c-kit in genesis, and yet another of the many emerging roles of the interstitial cell of Cajal in the pathogenesis of gastrointestinal diseases? Adv Anat Pathol. 1999 Jan;6(1):19-40. doi: 10.1097/00125480-199901000-00003. PMID 10197236
- [Result] Hirota S, Isozaki K, Moriyama Y, Hashimoto K, Nishida T, Ishiguro S, Kawano K, Hanada M, Kurata A, Takeda M, Muhammad Tunio G, Matsuzawa Y, Kanakura Y, Shinomura Y, Kitamura Y. Gain-of-function mutations of c-kit in human gastrointestinal stromal tumors. Science. 1998 Jan 23;279(5350):577-80. doi: 10.1126/science.279.5350.577. PMID 9438854
- [Result] Hirota S, Ohashi A, Nishida T, Isozaki K, Kinoshita K, Shinomura Y, Kitamura Y. Gain-of-function mutations of platelet-derived growth factor receptor alpha gene in gastrointestinal stromal tumors. Gastroenterology. 2003 Sep;125(3):660-7. doi: 10.1016/s0016-5085(03)01046-1. PMID 12949711
- [Result] Heinrich MC, Corless CL, Duensing A, McGreevey L, Chen CJ, Joseph N, Singer S, Griffith DJ, Haley A, Town A, Demetri GD, Fletcher CD, Fletcher JA. PDGFRA activating mutations in gastrointestinal stromal tumors. Science. 2003 Jan 31;299(5607):708-10. doi: 10.1126/science.1079666. Epub 2003 Jan 9. PMID 12522257
- [Result] Li J, Shen L. The current status of and prospects in research regarding gastrointestinal stromal tumors in China. Cancer. 2020 May 1;126 Suppl 9:2048-2053. doi: 10.1002/cncr.32684. PMID 32293728
- [Result] Cao F, Li A, Li J, Fang YU, Li F. Feasibility and safety of laparoscopic resection for gastric GISTs larger than 5 cm: Results from a prospective study. Oncol Lett. 2015 Oct;10(4):2081-2086. doi: 10.3892/ol.2015.3547. Epub 2015 Jul 30. PMID 26622800
- [Result] Huang CM, Chen QF, Lin JX, Lin M, Zheng CH, Li P, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Tu RH. Can laparoscopic surgery be applied in gastric gastrointestinal stromal tumors located in unfavorable sites?: A study based on the NCCN guidelines. Medicine (Baltimore). 2017 Apr;96(14):e6535. doi: 10.1097/MD.0000000000006535. PMID 28383420
- [Result] DeMatteo RP, Lewis JJ, Leung D, Mudan SS, Woodruff JM, Brennan MF. Two hundred gastrointestinal stromal tumors: recurrence patterns and prognostic factors for survival. Ann Surg. 2000 Jan;231(1):51-8. doi: 10.1097/00000658-200001000-00008. PMID 10636102
- [Result] Dematteo RP, Gold JS, Saran L, Gonen M, Liau KH, Maki RG, Singer S, Besmer P, Brennan MF, Antonescu CR. Tumor mitotic rate, size, and location independently predict recurrence after resection of primary gastrointestinal stromal tumor (GIST). Cancer. 2008 Feb 1;112(3):608-15. doi: 10.1002/cncr.23199. PMID 18076015
- [Result] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Result] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Result] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Result] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469